CLINICAL TRIAL: NCT02584023
Title: Preventive Effect of Lung Ultrasound and Alveolar Recruitment on Atelectasis in Mechanically Ventilated Infants
Brief Title: Lung Ultrasound and Alveolar Recruitment in Mechanically Ventilated Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-1509-063-703
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Atelectasis
Keywords: ultrasonography; infant; perioperative period; general anesthesia
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): No intervention during the perioperative period. Perform lung ultrasound twice only for the diagnostic purpose after the endotracheal intubation and and at the end of surgery.
  Interventions: Device: Lung ultrasound
- Alveolar recruitment (Active Comparator): Perform lung ultrasound twice during the perioperative period after the endotracheal intubation and and at the end of surgery. Conduct alveolar recruitment maneuver after first lung ultrasound assessment.
  Interventions: Device: Lung ultrasound

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasound on both hemithorax in supine position

SUMMARY:
Investigators hypothesized that lung ultrasound-assisted recruitment maneuver would be beneficial in mechanically ventilated infants compared to those who did not receive lung ultrasound and alveolar recruitment maneuver.

ELIGIBILITY:
Inclusion Criteria:

* Minor surgery less than 2 hours under general anesthesia
* Mechanically ventilated after endotracheal intubation

Exclusion Criteria:

* History of surgery on the lungs
* Laparoscopic surgery
* Abnormal preoperative chest radiograph findings including atelectasis, pneumothorax, pleural effusion, and pneumonia
* Considered inappropriate by the investigator

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postoperative incidence of pulmonary atelectasis | within the first day after the surgery

SECONDARY OUTCOMES:
Intraoperative incidence of pulmonary atelectasis after endotracheal intubation | from the moment of endotracheal intubation until the end of surgery, up to 6 hours
Intraoperative incidence of pulse oximetry (SpO2) ≤ 95% (or 10% below the baseline value) | from the induction of general anesthesia until the end of the surgery, up to 6 hours
Postoperative incidence of pulse oximetry (SpO2) ≤ 95% (or 10% below the baseline value) | within the first day after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Lutterbey G, Wattjes MP, Doerr D, Fischer NJ, Gieseke J Jr, Schild HH. Atelectasis in children undergoing either propofol infusion or positive pressure ventilation anesthesia for magnetic resonance imaging. Paediatr Anaesth. 2007 Feb;17(2):121-5. doi: 10.1111/j.1460-9592.2006.02045.x. PMID 17238882
- [Background] Magnusson L, Spahn DR. New concepts of atelectasis during general anaesthesia. Br J Anaesth. 2003 Jul;91(1):61-72. doi: 10.1093/bja/aeg085. No abstract available. PMID 12821566
- [Background] Tusman G, Bohm SH, Tempra A, Melkun F, Garcia E, Turchetto E, Mulder PG, Lachmann B. Effects of recruitment maneuver on atelectasis in anesthetized children. Anesthesiology. 2003 Jan;98(1):14-22. doi: 10.1097/00000542-200301000-00006. PMID 12502973
- [Background] Ashton-Cleary DT. Is thoracic ultrasound a viable alternative to conventional imaging in the critical care setting? Br J Anaesth. 2013 Aug;111(2):152-60. doi: 10.1093/bja/aet076. Epub 2013 Apr 12. PMID 23585400
- [Background] Kiley S, Cassara C, Fahy BG. Lung ultrasound in the intensive care unit. J Cardiothorac Vasc Anesth. 2015 Feb;29(1):196-203. doi: 10.1053/j.jvca.2014.10.017. No abstract available. PMID 25620145
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376